CLINICAL TRIAL: NCT04207723
Title: Effectiveness and Safety of Transcutaneous Posterior Tibial Nerve Stimulation for Premature Ejaculation Treatment
Brief Title: Transcutaneous Posterior Tibial Nerve Stimulation for Premature Ejaculation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMGC-5
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TENS Therapy (Experimental): Tens therapy + placebo drug therapy
  Interventions: Other: Transcutaneous posterior tibial nerve stimulation
- Control (Sham Comparator): Standard treatment (paroxetine 20 mg) + sham therapy
  Interventions: Drug: Paroxetine
- Combination therapy (Experimental): Tens therapy + standard treatment (paroxetine 20 mg)
  Interventions: Other: Transcutaneous posterior tibial nerve stimulation; Drug: Paroxetine

INTERVENTIONS:
Other: Transcutaneous posterior tibial nerve stimulation — Three (3) sessions per week per twelve (12) consecutive weeks, with a duration of 30 minutes each, with the application of 20 Hertz with a pulse amplitude of 200 MI sec. in each session. The intensity will be applied individually for each patient depending on the tolerance of the individual.
  Arms: Combination therapy; TENS Therapy
Drug: Paroxetine — paroxetine 20 mg / day taken in the morning hours, per 12 weeks.
  Arms: Combination therapy; Control

SUMMARY:
Objective: Evaluate the effectiveness and safety of transcutaneous electrostimulation of the posterior tibial nerve alone and combined with standard pharmacological treatment, in men with primary premature ejaculation, compared to standard pharmacological treatment.

Patients and methods: Randomized controlled clinical trial. Patients diagnosed with premature ejaculation attending Boston Medical Group clinics in Colombia and Spain will be included. Participants will be assigned by randomization to one of three treatment groups:

* Group 1: Tens + placebo drug therapy
* Group 2: Standard treatment (paroxetine 20 mg) + placebo therapy
* Group 3: Tens therapy + standard treatment (paroxetine mg)

The change in intravaginal latency time measured with the couple's sustained stopwatch, the change in the PEDT scale, the perception of the change in their initial condition after treatment (Global Clinical impression of change scale), and the change in different domains of the EP (PEP Scale - Profile Ejaculation Premature) at the end of treatment (week 12) and at three months of follow-up (week 24).

ELIGIBILITY:
Inclusion Criteria:

* Primary premature ejaculation as defined by the International Society for Sexual Medicine (ISSM-International Society for Sexual Medicine) (30): a) ejaculation occurs always or almost always within the first minute after penetration, b) disability to delay ejaculation in all or almost all penetrations, c) negative personal consequences are generated, such as stress, discomfort, frustration and / or avoidance of sexual intimacy.
* Age equal to or greater than 18 years.
* PEDT score greater than 11.
* Stable heterosexual relationship of at least 6 months with the interest of maintaining it for at least the duration of the study.
* Sexual activity at least once a week.
* Minimum chronicity of PE of 6 months.
* Voluntary participation in the study.
* Signature of informed consent prior to participation in the study.

Exclusion Criteria:

* IIEF-EF score greater than 25.
* Clinically significant comorbidity: cardiovascular, hepatic, thromboembolic, neurological, locomotive, endocrine, oncological, renal or rheumatologic.
* History of retroperitoneal surgery, radiotherapy or multiple sclerosis.
* History of mental illness: depression, anxiety, suicidal behavior, bipolar disorder, agoraphobia, dysthymia, social phobia, obsessive compulsive disorder, post-traumatic stress, psychiatric disorder, referred by the patient or by the use of a medication for one of these terms.
* Consumption of medications that affect ejaculatory control such as psychiatric medications, opioid analgesics, alpha blockers.
* Treatment for PD in the last 3 months.
* Treatment for epileptic syndromes or Parkinson's disease.
* Use of pacemaker or cardiac defibrillator.
* Skin lesions in the electrode placement area.
* Abuse or dependence on piscoactive substances: alcohol, hallucinogenic drugs.
* Couple in a state of pregnancy.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Intravaginal latency time at week 12 | Week 12
  Mean change in intravaginal latency time, measured with a stopwatch by the couple, at week 12.

SECONDARY OUTCOMES:
Change in Premature Ejaculation Diagnostic Tool (PEDT) questionnaire score | weeks 12 and 24
  Patients with a change in Premature Ejaculation Diagnostic Tool questionnaire score at weeks 12 and 24. A score of 11 or more suggests PE. A score of 9 or 10 may be found in men with PE; it is a "borderline" score. A score of 8 or less suggests that a man does not have PE. The minimum and maximum values are 0 and 20, respectively.
Clinical improvement | weeks 12 and 24
  Three-fold increase in intravaginal ejaculatory latency time

CONTACTS AND LOCATIONS:
Overall Officials: Héctor Corredor, Md, Principal Investigator — Boston Medical Group
Locations (1):
- Boston Medical Group, Bogotá, Bogota D.C., Colombia